CLINICAL TRIAL: NCT05886933
Title: A Prospective, Non-Intervention, Multi-Center Observational Study to Evaluate the Efficacy and Safety of FEXUCLUE Tablet in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Efficacy and Safety of FEXUCLUE Tablet
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWFE_P407
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fexuprazan Hydrochloride — Patient treated with Fexuprazan Hydrochloride (Fexuclue Tablet)
  Other Names: Fexuclue Tablet

SUMMARY:
This observational study is a large-scale, prospective, and multi-institutional observational study.

Patients from 19 to 75 years of age, will take a self-assessment (PRO) during the study period before and after administration of Pexuclue tablet.

DETAILED DESCRIPTION:
Data will be collected based on patient's medical records from daily visit. Enrolled subjects will take a Patient Reported Outcome (PRO) survey including Quality of life evaluation (GERD-HRQL) and self-awareness symptom (RDQ).

The survey will be done twice (before and after the administration of Fexuclue tablet) electronically through an application (e-PRO).

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 years to 75 years (on registration date)
2. Patient scheduled to administer Fexuclue tablet based on the medical judgment of investigator.
3. Patient who has not taken a treatment for gastroesophageal reflux disease within two weeks from baseline visit.
4. Patient who agreed to participate in this observation study and signed Informed Consent Form

Exclusion Criteria:

1. A person who falls under the prohibition of administration according to the permission for Fexuclue Tablet

   * Patients with hypersensitivity to the components of Fexuclue tablet or Fexuclue tablet and a history thereof
   * Patients undergoing Atazanavir, Nelfinavir or Lilpivirin-containing preparations
   * Pregnant and lactating women
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabortion
2. A person who has taken a treatment for gastroesophageal reflux disease within two weeks from baseline visit.
3. In addition to the above, a person who has determined that the researcher (the doctor in charge) is not suitable for participation in this observation study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referring to the minimum number of subjects required and the number of patients with gastroesophageal reflux disease in Korea, We expected to recruit about 16,000 people which is 0.2 %.
  However, since this study is conducted under daily medical care, we expected 10% to be dropout rate.
  Therefore the total study population is about 18,000
Sampling Method: Probability Sample
Enrollment: 9846 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the average score of the degree of individual symptoms of subjective symptoms (RDQ) | at least 4 weeks (up to 8 weeks)
  Average score change in Reflux Disease Questionnaire (0 ~5) from baseline
Change in the average score of the frequency of individual symptoms of subjective symptoms (RDQ) | at least 4 weeks (up to 8 weeks)
  Average score change in Reflux Disease Questionnaire (0 ~5) from baseline

SECONDARY OUTCOMES:
Changes in average score of the degree by symptoms (reflux, heartburn, indigestion) | at least 4 weeks (up to 8 weeks)
  Average score change in Reflux Disease Questionnaire (0 ~5) from baseline
Changes in average score of the frequency by symptoms (reflux, heartburn, indigestion) | at least 4 weeks (up to 8 weeks)
  Average score change in Reflux Disease Questionnaire (0 ~5) from baseline
RDQ validity rate | at least 4 weeks (up to 8 weeks)
  RDQ validity rate at 4 weeks(up to 8 weeks) from baseline
RDQ loss rate | at least 4 weeks (up to 8 weeks)
  RDQ loss rate at 4 weeks(up to 8 weeks) from baseline
Overall improvement evaluated by the subjects | at least 4 weeks (up to 8 weeks)
  Overall improvement result (scale 1~5, Fully recovered/Much improvement/Moderate improvement/Unchanged/Aggravated) evaluated by the subjects at 4 weeks(up to 8 weeks) from baseline
Overall improvement evaluated by the researchers | at least 4 weeks (up to 8 weeks)
  Overall improvement result (scale 1~5, Fully recovered/Much improvement/Moderate improvement/Unchanged/Aggravated) evaluated by the researchers at 4 weeks(up to 8 weeks) from baseline
Quality of Life (GERD-HRQL) Total score change | at least 4 weeks (up to 8 weeks)
  Quality of Life (GERD-HRQL) Total score change at 4 weeks(up to 8 weeks) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Homin Lee, Principal Investigator — Co&Ping Otolaryngology Clinic
Locations (1):
- Co&Ping Otolaryngology Clinic, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this point